CLINICAL TRIAL: NCT02465762
Title: Clinical Study to Evaluate the Safety and Efficacy of the UltraShape Device Using the U-Sculpt/VDF Transducer for Flanks Fat and Circumference Reduction
Brief Title: UltraShape Device Using the U-Sculpt/VDF Transducer for Flanks Fat
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Study design was amended to include a control - reregistered as NCT02465775
Sponsor: Syneron Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DHF18001
Record Dates: First submitted 2015-06-01; First posted 2015-06-08 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Unwanted Flanks Fat
Keywords: non-invasive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ultrashape fat reduction treatment (Experimental): all patient undergo non-invasive fat and circumference reduction at the flanks area
  Interventions: Device: ultrashape Fat reduction

INTERVENTIONS:
Device: ultrashape Fat reduction — Ultrashape Device focused ultrasound to produce localized mechanical motion within fat tissues and cells for the purpose of producing mechanical cellular membrane disruption. It is intended for reduction in abdominal circumference.
  Other Names: Ultrashape

SUMMARY:
Prospective, blinded, one arm, baseline-controlled clinical study for the evaluation of the UltraShape treatment for non-invasive fat and circumference reduction.

Study subjects will undergo UltraShape treatments on the flanks area using the U-Sculpt/VDF Transducer - 60 subjects.

DETAILED DESCRIPTION:
This study is a prospective, baseline and blinded controlled, one arm clinical study showing the performance and safety of the UltraShape treatment for non-invasive fat and circumference reduction at the flanks area.

Up to 60 Healthy subjects in up to 4 investigational sites will be enrolled in this study. All subjects will undergo an assessment of their general health. During the treatment period, subject's circumference and fat thickness will be measured and three successive bi-weekly (two weeks interval) UltraShape treatments will be performed.

The study subjects will undergo UltraShape treatments on the flanks area using the U-Sculpt /VDF Transducer.

During the follow-up period visit will be conducted as follow: 4 weeks (4wk FU), 8 weeks (8wk FU) and 16 weeks (16wk FU) post last treatment (Tx.3). Subject's circumference will be measured in the measurements points according to the flanks treated area, circumference reduction will be assessed at each visit. Additionally, a subject questionnaire will be completed in each follow-up visit. Finally, photography will be performed under visible light conditions of the front, right, left and back view. Most of the assessments will occur at each of the visits to the clinic.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent to participate in the study.
2. Female and male subjects, between 18 to 60 years of age at the time of enrolment
3. Fitzpatrick Skin Type I to VI.
4. Fat thickness of at least 1.5 cm in the treated area (measured by calibrated caliper).
5. BMI interval: BMI between 22 to 30 (normal to overweight, but not obese).
6. If female, not pregnant or lactating, must be either post-menopausal, surgically sterilized, or using a medically acceptable form of birth control at least 3 months prior to enrollment (i.e., oral contraceptives, contraceptive implant, barrier methods with spermicide or abstinence).
7. In addition, negative urine pregnancy test as tested before each treatment and at the last follow-up visit for women with child-bearing potential (e.g. not menopause).
8. General good health confirmed by medical history and skin examination of the treated area.
9. Willing to follow the treatment and follow-up schedule and post-treatment care instructions.
10. Willingness to refrain from a change in diet/ exercise/medication regimen for the entire course of the study.
11. Willing to have photographs and images taken of the treated areas to be used, de-identified in evaluations, publications and presentations.

Exclusion Criteria:

1. History of hypertension, ischemic heart disease, valvular heart disease, congestive heart failure, pacemaker/defibrillator, abdominal aortic aneurism
2. Known hyperlipidemia, diabetes mellitus, hepatitis, liver disease, HIV positive status, blood coagulopathy or excessive bleeding, autoimmune or connective tissue disease
3. Having or undergoing any form of treatment for active cancer, or having a history of skin cancer or any other cancer in the areas to be treated, including presence of malignant or pre-malignant pigmented lesions
4. Having any active electrical implant anywhere in the body, such as a pacemaker or an internal defibrillator
5. Having a permanent implant in the treated area, such as metal plates or an injected chemical substance such as silicone
6. Having undergone any other surgery in the treated areas within 12 months of treatment or during the study, including liposuction
7. Previous body contouring procedures in the treatment area within 12 months
8. History of skin disease in the treatment area, known tendency to form keloids or poor wound healing
9. Suffering from significant skin conditions in the treated areas or inflammatory skin conditions, including, but not limited to, open lacerations or abrasions and active cold sores or herpes sores prior to treatment (duration of resolution as per the Investigator's discretion) or during the treatment course
10. Skin lesions in the treatment area other than simple nevi on physical examination (e.g., atypical nevus, tattoo, abrasions) including depressed scars in the treatment area
11. Very poor skin quality (i.e., severe laxity)
12. Abdominal wall diastasis or hernia on physical examination
13. Abnormal kidney, liver or coagulation functions, abnormal lipid profile or blood count within the last 3 months
14. Obesity (BMI above 30)
15. Childbirth within the last 12 months or breastfeeding women. Any acute or chronic condition which, in the opinion of the investigator, could interfere with the conduct of the study
16. Unstable weight within the last 6 months (i.e., ± 3% weight change in the prior six months)
17. Inability to comply with circumference measurement procedure (e.g., inability to hold breath for the required duration).
18. Fat thickness lower than 2.5 cm after strapping at the treated area.
19. Participation in another clinical study involving same anatomical areas within the last 6 months (or 30 days in case different anatomical areas were treated in previous trial/s).
20. As per the Investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-08; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Efficacy flanks fat reduction | 4, 8 and 16 weeks post last treatment (Tx.3)
  measure by caliper and Ultrasound

SECONDARY OUTCOMES:
circumference reduction post UltraShape treatments | 4, 8 and 16 weeks post last treatment (Tx.3)
  Reduction will be calculated
fat thickness reduction | 4, 8 and 16 weeks post last treatment (Tx.3)
  by caliper and by Ultrasound device
Investigator satisfaction assessment | 4, 8 and 16 weeks post last treatment (Tx.3)
  5-Point Likert Scale
Subject satisfaction assessment | 4, 8 and 16 weeks post last treatment (Tx.3)
  The subjects will answer the questionnaire
Comfort level | day 0, after 2 and 4 weeks
  using NSR scale
Evaluate the safety for flanks fat reduction | up to 20 weeks
  Evaluate the safety of the treatment with the UltraShape device using the U-Sculpt/VDF Transducer for flanks treatment area

CONTACTS AND LOCATIONS:
Overall Officials: William P Coleman, MD, Principal Investigator — Coleman Center for Cosmetic Dermatologic Surgery 4425 Conlin Street, Metairie, Louisiana 70006; Michael Gold, MD, Principal Investigator — Gold Skin Care Center, 2000 Richard Jones Road, Suite 220, Nashville, TN 37215 USA; Robert Weiss, MD, Principal Investigator — 54 Scot Adams Road, Hunt Valley Baltimore USA

REFERENCES:
- [Background] Adamo C, Mazzocchi M, Rossi A, Scuderi N. Ultrasonic liposculpturing: extrapolations from the analysis of in vivo sonicated adipose tissue. Plast Reconstr Surg. 1997 Jul;100(1):220-6. doi: 10.1097/00006534-199707000-00033. PMID 9207679
- [Background] Goldman A. Submental Nd:Yag laser-assisted liposuction. Lasers Surg Med. 2006 Mar;38(3):181-4. doi: 10.1002/lsm.20270. PMID 16453321
- [Background] Hexsel D, Serra M, Mazzuco R, Dal'Forno T, Zechmeister D. Phosphatidylcholine in the treatment of localized fat. J Drugs Dermatol. 2003 Oct;2(5):511-8. PMID 14558399